CLINICAL TRIAL: NCT06428838
Title: Eptinezumab as an Adjunct to Standard of Care for MIGRANE in an Acute EmeRgency Context (Migraine ERase Study)
Brief Title: Eptinezumab as an Adjunct to Standard of Care for Migraine in an Acute Emergency Context
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr George Medvedev (Industry)
Collaborators: H. Lundbeck A/S (Industry); Centre for Neurology Studies, Surrey Neuroplasticity Clinic Inc. (Unknown); Royal Columbian Hospital Foundation (Other); Surrey Memorial Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Dr George Medvedev, Principal Investigator, HealthTech Connex Inc.
Organization: HealthTech Connex Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Medvedev_001
Record Dates: First submitted 2024-05-16; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Migraine; Chronic Migraine
Keywords: acute treatment; emergency; monoclonal antibody
MeSH Terms: conditions — Migraine Disorders; Emergencies | interventions — eptinezumab; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized (1:1), controlled trial with standard of care (SoC) as control arm.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Other): SoC will be delivered at the discretion of the treating physician
  Interventions: Other: Standard of Care
- Standard of Care + Eptinezumab (Experimental): In addition to standard of care, participants randomized to the Standard of Care + Eptinezumab arm will receive a single infusion of eptinezumab (100mg/mL).
  Interventions: Biological: Eptinezumab; Other: Standard of Care

INTERVENTIONS:
Biological: Eptinezumab — The study treatment consists of a single infusion of eptinezumab (100mg/mL).
  Arms: Standard of Care + Eptinezumab
Other: Standard of Care — SoC may include a combination of Toradol, Metoclopramide, and/or Benadryl. Ketamine and/or Midazolam may also be used, according to a stepwise approach, at the discretion of the treating physician. The timing and dose of all medication(s) administered in the ED will be recorded.

SUMMARY:
The purpose of the study is to investigate how a medication called eptinezumab (Vyepti) given to patients in the Emergency Department (ED) might help prevent migraines from happening again. The results of this study may help inform better ways to manage patients with migraines in the ED.

Eptinezumab is currently approved by Health Canada for the preventive treatment of migraine, but its short-term effectiveness in the ED context is unknown. Unlike other migraine treatments used in the ED, eptinezumab can rapidly interrupt the migraine process, potentially also preventing migraine from coming back in the short term.

Most patients with a diagnosis of migraine have no access to preventative therapies. This study will be able to provide access to preventative therapy at the earliest stages of a migraine attack. Administering this medication in the ED may stop the attack more effectively compared to current therapies.

This study wants to see if eptinezumab could help stop migraines from coming back after individuals have been treated in the ED. The study will also explore whether eptinezumab could reduce how often individuals with migraine might need to come back to the ED, what other medications they might need alongside eptinezumab, and how they feel overall.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between the ages of 19-75 with a history of migraines, as established at the time of presentation to the ED or known from the patient's chart;
2. Presenting to the emergency department with a migraine that meets ICHD-3 migraine headache criteria;
3. Provided signed informed consent;
4. Sufficient literacy and cognitive capacity to understand and complete patient self-rated questionnaires in English.

Exclusion Criteria:

1. Secondary headaches caused by an injury or underlying illness, such as a concussion, bleeding in the brain, an infection or a brain tumor
2. Current or history of severe cardiovascular disease or renal dysfunction
3. A systemic condition in the stage of active treatment (vasculitis, etc.)
4. Pregnant or at risk of becoming pregnant (absent contraception)
5. Currently enrolled in another investigational drug trial
6. Dosed with eptinezumab within the past 3 months
7. Currently on anti-CGRP therapy with monoclonal antibodies
8. Currently involved in active litigation
9. Any other condition which, in the opinion of the Investigator, would exclude the participant due to reasons of safety or data integrity
10. Hypersensitivity to the active substance or to any of the excipients

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of migraine days at week 1 | Baseline to Week 1
  Number of migraine days at week 1, as reported in daily Headache Diary

SECONDARY OUTCOMES:
Readmission to the Emergency Department (ED) | Baseline to Month 3
  Readmission to the Emergency Department (ED) as assessed by patient chart
Generalized Anxiety Disorder 7-item (GAD-7) | Baseline to Month 3
  The Generalized Anxiety Disorder 7-item (GAD-7) will be assessed at baseline, month 1 and month 3. The GAD-7 is a short self-report questionnaire assessing the severity of anxiety disorder. For each item, the participant is asked how bothered they have been by the problem in the last 2 weeks. The total score ranges from 0-21, and a score greater than 15 indicates severe anxiety. The recall period for the GAD-7 is 2 weeks.
Headache Impact Test (HIT-6) | Baseline to Month 3
  The Headache Impact Test (HIT-6) will involve an assessment at baseline and at months 1 and 3. The HIT-6 (v1.0) is a Likert-type, self-reported questionnaire designed to assess the impact of an occurring headache and its effect on the ability to function normally in daily life. HIT-6 scores range from 36 to 78. Higher scores indicate a greater impact of headaches on the respondent's life, i.e., 36 = no impact, 78 = maximum impact. The HIT-6 consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. The assessment was developed to measure a wide spectrum of factors contributing to headache burden, and it has demonstrated reliability and validity. The recall period for the HIT-6 is 4 weeks.
Patient Health Questionnaire (PHQ-9) | Baseline to Month 3
  The PHQ-9 is a short self-report questionnaire assessing signs and symptoms of depression. The questionnaire consists of nine items which ask about the frequency and severity of depressive symptoms based on DSM-IV criteria. For each item, the participant is asked to rate the severity of the symptom on a scale from 0 to 3. The total score ranges from 0-27 with a higher score indicating more severe depressive symptoms. The recall period for the PHQ-9 is 2 weeks.
Patient Global Impression of Change (PGI-C) | Baseline to Month 3
  The PGI-C will involve an assessment at 24-72hrs, week 1, month 1 and month 3. PGI-C is a one-item measure rating of the overall patient perceived improvement on a seven-point scale. Patients rate their change since treatment initiation as "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse", or "very much worse.
Number of monthly headache days | Baseline to Month 3
  Number of monthly headache days as assessed by the Migraine Disability Assessment (MIDAS)
Migraine recurrence | Baseline to Month 3
  Recurrence of migraine as reported in daily Headache Diary
Work Productivity and Activity Impairment (WPAI) | Baseline to Month 3
  The WPAI is a six-item validated instrument that measures aspects of work productivity and activity impairment due to migraine over the past 7 days with higher values, in the form of percentages, indicating greater impairment due to the respondent's health. Only patients that are currently employed (full-time, part-time, or self-employed) are eligible to respond to the items assessing work-related activities. Item 6 in the WPAI will be administered to those not in employment, providing the possibility of calculating activity impairment for patients that are not employed. The six items are used to derive four subscales: Absenteeism (proportion of missed work hours out of the total; scale 0-100%), Presenteeism (level of work impairment; scale 0-10), Overall work impairment (combination of absenteeism and presenteeism; scale 0-100%), and Activity impairment (impairment in daily activities; scale 0-10).
Sleep Quality | Baseline to Month 3
  Sleep quality will be assessed with the question, "On average, about how many hours of sleep do you get per night?" with responses including "7-9 hrs", "6-6.9 hrs", "5-5.9 hrs" or "less than 5 hrs". The recall period will be 1 week.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia

IPD SHARING:
Plan to Share IPD: No
If the results of the study are published in the public domain, only aggregate/group data will be published.